CLINICAL TRIAL: NCT00884117
Title: Influenza Resistance Information Study (IRIS)
Brief Title: Influenza Resistance Information Study
Acronym: IRIS
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: NV20237; 2008-006149-24 (EudraCT Number)
Record Dates: First submitted 2009-04-15; First posted 2009-04-20 (Estimated); Results first posted 2016-07-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Participants Infected with Influenza: Participants with a positive diagnostic test of influenza and/or displaying symptoms suggestive of influenza-like illness will be enrolled and followed for up to 10 days after informed consent for virological surveillance and assessment of clinical outcomes. Participants may receive treatment including oseltamivir, other treatment/medication, or no treatment.
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Oseltamivir — Participants may receive treatment at the discretion of the investigator according to local practice standards, and there is no protocol-specified intervention. However, analyses will be presented separately for participants treated with oseltamivir during the course of the study.
  Other Names: Tamiflu

SUMMARY:
This study will assist in the early detection of influenza resistant to antivirals and will monitor the clinical outcome of adults and children infected with influenza according to subtype and susceptibility. Participants clinically diagnosed with influenza will undergo a rapid diagnostic test and viral sampling at Baseline and on Days 3, 6, and 10. Participants will be clinically managed according to local guidelines and the decision to treat/not treat will be at the discretion of the Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Participants greater than or equal to (≥) 1 year of age with a positive diagnostic test of influenza and/or displaying symptoms suggestive of influenza-like illness (during Years 1 to 5)
* Participants less than or equal to (≤) 12 years of age with a positive diagnostic test of influenza and displaying symptoms suggestive of influenza-like illness and who are being or, according to local standard of care, will be treated with an influenza antiviral (during Years 6 and 7)

Exclusion Criteria:

* Allergy to any potential influenza therapy
* Living in the same household or residential/care home as another study participant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with a positive diagnostic test of influenza and/or displaying symptoms suggestive of influenza-like illness will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 4561 (Actual)
Dates: Start 2009-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- Chicago, Illinois, United States
- Westmead, New South Wales, Australia
- Bron, France
- Berlin, Germany
- Shatin, Hong Kong
- Rotterdam, Netherlands
- Sandnes, Norway
- Krakow, Poland

REFERENCES:
- [Derived] Roosenhoff R, Reed V, Kenwright A, Schutten M, Boucher CA, Monto A, Clinch B, Kumar D, Whitley R, Nguyen-Van-Tam JS, Osterhaus ADME, Fouchier RAM, Fraaij PLA. Viral Kinetics and Resistance Development in Children Treated with Neuraminidase Inhibitors: The Influenza Resistance Information Study (IRIS). Clin Infect Dis. 2020 Aug 22;71(5):1186-1194. doi: 10.1093/cid/ciz939. PMID 31560055
- [Derived] Fraaij PL, Schutten M, Javouhey E, Burleigh L, Outlaw R, Kumar D, Boucher CA. Viral shedding and susceptibility to oseltamivir in hospitalized immunocompromised patients with influenza in the Influenza Resistance Information Study (IRIS). Antivir Ther. 2015;20(6):633-42. doi: 10.3851/IMP2957. Epub 2015 Apr 7. PMID 25849228

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants Infected With Influenza: Participants with a positive diagnostic test of influenza and/or displaying symptoms suggestive of influenza-like illness were enrolled. During Years 1 to 5 of the overall study, otherwise healthy/non-immunocompromised adults and children greater than or equal to (≥) 1 year of age were considered as eligible. Following a protocol amendment, inclusion criteria for Years 6 and 7 were changed to only include healthy or immunocompromised children less than or equal to (≤) 12 years of age being treated with an influenza antiviral medication. Participants were followed for up to 10 days after informed consent for virological surveillance and assessment of clinical outcomes.
Period: Overall Study
Arm/Group | All Participants Infected With Influenza
Started | 4561
Completed | 4312 (Defined as Day 6 visit for those enrolled before Amendment D; thereafter defined as Day 10 visit.)
Not Completed | 249
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 89
Not completed — Death | 3
Not completed — Lost to Follow-up | 143
Not completed — Other | 12

BASELINE CHARACTERISTICS:
Population: All Enrolled Healthy Participants (AEHP) Population: All otherwise healthy participants who entered the study. Due to the imbalance between healthy (n=4553) and immunocompromised participants (n=8), results from immunocompromised participants were not included in any analyses, and data obtained from healthy participants were the focus of the study.
Groups:
- Otherwise Healthy Participants Infected With Influenza: Otherwise healthy/non-immunocompromised participants with a positive diagnostic test of influenza and/or displaying symptoms suggestive of influenza-like illness were enrolled. During Years 1 to 5 of the overall study, adults and children ≥1 year of age were considered as eligible. Following a protocol amendment, inclusion criteria for Years 6 and 7 were changed to only include children ≤12 years of age being treated with an influenza antiviral medication. Participants were followed for up to 10 days after informed consent for virological surveillance and assessment of clinical outcomes.
Arm/Group | Otherwise Healthy Participants Infected With Influenza
Number analyzed (Participants) | 4553
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.5 (19.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2331
  Male | 2222

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Genotypic Resistance
Description: Samples were analyzed using reverse transcriptase-polymerase chain reaction (RT-PCR). Pre-defined mutations in viral ribonucleic acid (RNA) were noted, the presence of which was defined as genotypic resistance. The number of participants with genotypic resistance at Baseline was reported. The number of participants with genotypic resistance post-Baseline was determined by a collective count of all participants who had a resistance mutation at least once on Days 3, 6, and/or 10. (Hereafter, "H" stands for hemagglutinin and "N" stands for neuraminidase in abbreviations of viral subtype such as H1N1, H1N1pdm09, and H3N2.)
Time Frame: Baseline (Day 1) and post-Baseline (Days 3, 6, 10)
Population: All Laboratory-Confirmed Influenza Participants (ALCIP) Population: All with confirmed influenza by positive RT-PCR at Baseline. The "Number of Participants Analyzed" reflects the total of participants who provided evaluable data for their viral RNA subtype. The number who provided data for each viral RNA subtype in each timeframe (n) is shown.
Measure: Number; unit: participants
Arm/Group | Otherwise Healthy Participants Infected With Influenza
Number analyzed (Participants) | 3725
participants
  Baseline, H1N1 Seasonal (n=47) | 44
  Baseline, H1N1pdm09 (n=1240) | 1
  Baseline, H3N2 (n=1432) | 0
  Baseline, Influenza B (n=1006) | 2
  Baseline, All Types/Subtypes (n=3725) | 47
  Post-Baseline, H1N1 Seasonal (n=47) | 0
  Post-Baseline, H1N1pdm09 (n=1240) | 39
  Post-Baseline, H3N2 (n=1432) | 18
  Post-Baseline, Influenza B (n=1006) | 0
  Post-Baseline, All Types/Subtypes (n=3725) | 57

2. Primary Outcome: Percentage of Participants Exhibiting Treatment-Emergent Resistance by Study Year Among Participants With H3N2 or H1N1pdm09 Infections
Description: Pre-defined mutations in viral RNA were noted, the presence of which was defined as genotypic resistance. Treatment-emergent resistance was defined as the presence of genotypic or phenotypic resistance from a post-Baseline sample in the setting of a previously non-resistant Baseline sample. The percentage of participants with treatment-emergent resistance was reported by study year for participants with H3N2 or H1N1pdm09 infections. Only data with evaluable participants were reported.
Time Frame: From Baseline (Day 1) to Day 10 (assessed on Days 1, 3, 6, 10) during Study Years 1, 2, 3, 4, 5, 6, 7
Population: ALCIP Population. The "Number of Participants Analyzed" reflects combined H3N2 or H1N1pdm09-infected participants across all study years who provided an analyzable post-Baseline sample for their viral RNA subtype. The number of participants who provided evaluable data for each viral RNA subtype in the specified timeframe (n) is shown in the table.
Measure: Number; unit: percentage of participants
Groups:
- Children <1 Year of Age Treated With Oseltamivir: Otherwise healthy/non-immunocompromised children less than (<) 1 year of age with a positive diagnostic test of influenza and/or displaying symptoms suggestive of influenza-like illness were enrolled during Years 6 and 7 of the overall study. Participants receiving antiviral treatment with oseltamivir (according to local practice standards) were followed for up to 10 days after informed consent for virological surveillance and assessment of clinical outcomes.
- Children 1 to 5 Years of Age Treated With Oseltamivir: Otherwise healthy/non-immunocompromised children 1 to 5 years of age with a positive diagnostic test of influenza and/or displaying symptoms suggestive of influenza-like illness were enrolled during Years 1 to 7 of the overall study. Participants receiving antiviral treatment with oseltamivir (according to local practice standards) were followed for up to 10 days after informed consent for virological surveillance and assessment of clinical outcomes.
- Children 6 to 12 Years of Age Treated With Oseltamivir: Otherwise healthy/non-immunocompromised children 6 to 12 years of age with a positive diagnostic test of influenza and/or displaying symptoms suggestive of influenza-like illness were enrolled during Years 1 to 7 of the overall study. Participants receiving antiviral treatment with oseltamivir (according to local practice standards) were followed for up to 10 days after informed consent for virological surveillance and assessment of clinical outcomes.
- Children Treated With Oseltamivir: Otherwise healthy/non-immunocompromised children with a positive diagnostic test of influenza and/or displaying symptoms suggestive of influenza-like illness were enrolled during Years 1 to 7 of the overall study. Participants receiving antiviral treatment with oseltamivir (according to local practice standards) were followed for up to 10 days after informed consent for virological surveillance and assessment of clinical outcomes.
- Adults Treated With Oseltamivir: Otherwise healthy/non-immunocompromised adults with a positive diagnostic test of influenza and/or displaying symptoms suggestive of influenza-like illness were enrolled during Years 1 to 5 of the overall study. Participants receiving antiviral treatment with oseltamivir (according to local practice standards) were followed for up to 10 days after informed consent for virological surveillance and assessment of clinical outcomes.
- Participants Treated With Oseltamivir: Otherwise healthy/non-immunocompromised adults and children with a positive diagnostic test of influenza and/or displaying symptoms suggestive of influenza-like illness were enrolled during Years 1 to 7 of the overall study. Participants receiving antiviral treatment with oseltamivir (according to local practice standards) were followed for up to 10 days after informed consent for virological surveillance and assessment of clinical outcomes.
Arm/Group | Children <1 Year of Age Treated With Oseltamivir | Children 1 to 5 Years of Age Treated With Oseltamivir | Children 6 to 12 Years of Age Treated With Oseltamivir | Children Treated With Oseltamivir | Adults Treated With Oseltamivir | Participants Treated With Oseltamivir
Number analyzed (Participants) | 20 | 473 | 438 | 931 | 713 | 1644
percentage of participants
  Year 1, H3N2 (n=0,1,1,2,2,4) | NA — No participants were included in the analysis. | 0 | 0 | 0 | 0 | 0
  Year 2, H1N1pdm09 (n=0,54,81,135,108,243) | NA — No participants were included in the analysis. | 1.9 | 0 | 0.7 | 0.9 | 0.8
  Year 2, H3N2 (n=0,0,0,0,22,22) | NA — No participants were included in the analysis. | NA — No participants were included in the analysis. | NA — No participants were included in the analysis. | NA — No participants were included in the analysis. | 0 | 0
  Year 3, H1N1pdm09 (n=0,58,30,88,148,236) | NA — No participants were included in the analysis. | 20.7 | 3.3 | 14.8 | 1.4 | 6.4
  Year 3, H3N2 (n=0,37,43,80,122,202) | NA — No participants were included in the analysis. | 2.7 | 0 | 1.3 | 0.8 | 1.0
  Year 4, H1N1pdm09 (n=0,6,6,12,16,28) | NA — No participants were included in the analysis. | 16.7 | 0 | 8.3 | 0 | 3.6
  Year 4, H3N2 (n=0,19,17,36,67,103) | NA — No participants were included in the analysis. | 10.5 | 11.8 | 11.1 | 0 | 3.9
  Year 5, H1N1pdm09 (n=0,29,8,37,41,78) | NA — No participants were included in the analysis. | 20.7 | 12.5 | 18.9 | 4.9 | 11.5
  Year 5, H3N2 (n=0,82,80,162,187,349) | NA — No participants were included in the analysis. | 8.5 | 1.3 | 4.9 | 1.1 | 2.9
  Year 6, H1N1pdm09 (n=11,33,25,69,0,69) | 36.4 | 6.1 | 4.0 | 10.1 | NA — No participants were included in the analysis. | 10.1
  Year 6, H3N2 (n=1,45,27,73,0,73) | 0 | 0 | 0 | 0 | NA — No participants were included in the analysis. | 0
  Year 7, H1N1pdm09 (n=0,15,5,20,0,20) | NA — No participants were included in the analysis. | 33.3 | 0 | 25.0 | NA — No participants were included in the analysis. | 25.0
  Year 7, H3N2 (n=8,94,115,217,0,217) | 0 | 1.1 | 0.9 | 0.9 | NA — No participants were included in the analysis. | 0.9

3. Secondary Outcome: Number of Participants With Viral RNA Detected by RT-PCR on Day 1 Among Adults Treated With Oseltamivir
Time Frame: Baseline (Day 1)
Population: ALCIP Population. The "Number of Participants Analyzed" reflects the total number of participants who provided evaluable data for their viral RNA subtype at the Baseline visit.
Measure: Number; unit: participants
Arm/Group | Adults Treated With Oseltamivir
Number analyzed (Participants) | 961
participants
  Total | 961
  H1N1 Seasonal | 12
  H3N2 | 419
  H1N1pdm09 | 323
  Influenza B | 207

4. Secondary Outcome: Number of Participants With Viral RNA Detected by RT-PCR on Day 3 Among Adults Treated With Oseltamivir
Time Frame: Day 3
Population: ALCIP Population. The "Number of Participants Analyzed" reflects the total number of participants who provided evaluable data for their viral RNA subtype at the Day 3 visit. The number of participants who provided evaluable data for each viral RNA subtype at the Day 3 visit (n) is shown in the table.
Measure: Number; unit: participants
Arm/Group | Adults Treated With Oseltamivir
Number analyzed (Participants) | 912
participants
  Total (n=912) | 781
  H1N1 Seasonal (n=11) | 10
  H3N2 (n=398) | 341
  H1N1pdm09 (n=308) | 258
  Influenza B (n=195) | 172

5. Secondary Outcome: Number of Participants With Viral RNA Detected by RT-PCR on Day 6 Among Adults Treated With Oseltamivir
Time Frame: Day 6
Population: ALCIP Population. The "Number of Participants Analyzed" reflects the total number of participants who provided evaluable data for their viral RNA subtype at the Day 6 visit. The number of participants who provided evaluable data for each viral RNA subtype at the Day 6 visit (n) is shown in the table.
Measure: Number; unit: participants
Arm/Group | Adults Treated With Oseltamivir
Number analyzed (Participants) | 889
participants
  Total (n=889) | 317
  H1N1 Seasonal (n=9) | 4
  H3N2 (n=382) | 144
  H1N1pdm09 (n=308) | 110
  Influenza B (n=190) | 59

6. Secondary Outcome: Number of Participants With Viral RNA Detected by RT-PCR on Day 10 Among Adults Treated With Oseltamivir
Time Frame: Day 10
Population: ALCIP Population. The "Number of Participants Analyzed" reflects the total number of participants who provided evaluable data for their viral RNA subtype at the Day 10 visit. The number of participants who provided evaluable data for each viral RNA subtype at the Day 10 visit (n) is shown in the table.
Measure: Number; unit: participants
Arm/Group | Adults Treated With Oseltamivir
Number analyzed (Participants) | 833
participants
  Total (n=833) | 88
  H3N2 (n=362) | 44
  H1N1pdm09 (n=283) | 33
  Influenza B (n=188) | 11

7. Secondary Outcome: Number of Participants With Viral RNA Detected by RT-PCR on Day 1 Among Children Treated With Oseltamivir
Time Frame: Baseline (Day 1)
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Children Treated With Oseltamivir
Number analyzed (Participants) | 1283
participants
  Total | 1283
  H3N2 | 583
  H1N1pdm09 | 371
  Influenza B | 329

8. Secondary Outcome: Number of Participants With Viral RNA Detected by RT-PCR on Day 3 Among Children Treated With Oseltamivir
Time Frame: Day 3
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Children Treated With Oseltamivir
Number analyzed (Participants) | 1238
participants
  Total (n=1238) | 1050
  H3N2 (n=562) | 453
  H1N1pdm09 (n=358) | 315
  Influenza B (n=318) | 282

9. Secondary Outcome: Number of Participants With Viral RNA Detected by RT-PCR on Day 6 Among Children Treated With Oseltamivir
Time Frame: Day 6
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Children Treated With Oseltamivir
Number analyzed (Participants) | 1250
participants
  Total (n=1250) | 628
  H3N2 (n=567) | 271
  H1N1pdm09 (n=362) | 181
  Influenza B (n=321) | 176

10. Secondary Outcome: Number of Participants With Viral RNA Detected by RT-PCR on Day 10 Among Children Treated With Oseltamivir
Time Frame: Day 10
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Children Treated With Oseltamivir
Number analyzed (Participants) | 1228
participants
  Total (n=1228) | 197
  H3N2 (n=560) | 73
  H1N1pdm09 (n=351) | 64
  Influenza B (n=317) | 60

11. Secondary Outcome: Time to Non-Detection of Viral RNA
Description: Time to non-detection/viral clearance was the time between symptom onset and the day on which viral RNA was no longer detected, or the last visit date if the participant was not RNA-negative at that visit. Time to non-detection/viral clearance was estimated using Kaplan-Meier analysis and expressed in days.
Time Frame: From Baseline (Day 1) to Day 10 (assessed on Days 1, 3, 6, 10)
Population: ALCIP Population. The "Number of Participants Analyzed" reflects the number of participants who provided sufficient post-Baseline data.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Children ≤5 Years of Age Treated With Oseltamivir: Otherwise healthy/non-immunocompromised children ≤5 years of age with a positive diagnostic test of influenza and/or displaying symptoms suggestive of influenza-like illness were enrolled during Years 1 to 7 of the overall study. Participants receiving antiviral treatment with oseltamivir (according to local practice standards) were followed for up to 10 days after informed consent for virological surveillance and assessment of clinical outcomes.
Arm/Group | Children ≤5 Years of Age Treated With Oseltamivir | Children 6 to 12 Years of Age Treated With Oseltamivir | Adults Treated With Oseltamivir
Number analyzed (Participants) | 637 | 644 | 949
days | 9.7 [9.3 to 9.9] | 8.2 [8.0 to 9.1] | 7.9 [7.6 to 8.1]
Statistical Analysis 1: Comparison: Children ≤5 Years of Age Treated With Oseltamivir vs Children 6 to 12 Years of Age Treated With Oseltamivir vs Adults Treated With Oseltamivir; Test type: Superiority or Other; p < 0.0001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Children ≤5 Years of Age Treated With Oseltamivir vs Children 6 to 12 Years of Age Treated With Oseltamivir; Test type: Superiority or Other; p < 0.01, Pairwise Wilcoxon
Statistical Analysis 3: Comparison: Children ≤5 Years of Age Treated With Oseltamivir vs Adults Treated With Oseltamivir; Test type: Superiority or Other; p < 0.01, Pairwise Wilcoxon

12. Secondary Outcome: Time to Non-Detection of Viral RNA Among Participants With H3N2 Infections
Description: as for outcome 11
Time Frame: From Baseline (Day 1) to Day 10 (assessed on Days 1, 3, 6, 10)
Population: ALCIP Population. The "Number of Participants Analyzed" reflects the number of participants with H3N2 infection who provided sufficient post-Baseline data.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Children ≤5 Years of Age Treated With Oseltamivir | Children 6 to 12 Years of Age Treated With Oseltamivir | Adults Treated With Oseltamivir
Number analyzed (Participants) | 295 | 287 | 419
days | 9.5 [8.6 to 10.0] | 8.0 [7.1 to 8.7] | 8.0 [7.7 to 8.5]
Statistical Analysis 1: Comparison: Children ≤5 Years of Age Treated With Oseltamivir vs Children 6 to 12 Years of Age Treated With Oseltamivir vs Adults Treated With Oseltamivir; Test type: Superiority or Other; p = 0.015, Kruskal-Wallis
Statistical Analysis 2: Comparison: Children ≤5 Years of Age Treated With Oseltamivir vs Children 6 to 12 Years of Age Treated With Oseltamivir; Test type: Superiority or Other; p = 0.009, Pairwise Wilcoxon
Statistical Analysis 3: Comparison: Children 6 to 12 Years of Age Treated With Oseltamivir vs Adults Treated With Oseltamivir; Test type: Superiority or Other; p = 0.03, Pairwise Wilcoxon

13. Secondary Outcome: Time to Non-Detection of Viral RNA Among Participants With H1N1pdm09 Infections
Description: as for outcome 11
Time Frame: From Baseline (Day 1) to Day 10 (assessed on Days 1, 3, 6, 10)
Population: ALCIP Population. The "Number of Participants Analyzed" reflects the number of participants with H1N1pdm09 infection who provided sufficient post-Baseline data.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Children ≤5 Years of Age Treated With Oseltamivir | Children 6 to 12 Years of Age Treated With Oseltamivir | Adults Treated With Oseltamivir
Number analyzed (Participants) | 212 | 158 | 323
days | 9.9 [9.5 to 10.2] | 8.0 [7.0 to 8.9] | 8.0 [7.4 to 8.2]
Statistical Analysis 1: Comparison: Children ≤5 Years of Age Treated With Oseltamivir vs Children 6 to 12 Years of Age Treated With Oseltamivir vs Adults Treated With Oseltamivir; Test type: Superiority or Other; p = 0.0005, Kruskal-Wallis
Statistical Analysis 2: Comparison: Children ≤5 Years of Age Treated With Oseltamivir vs Children 6 to 12 Years of Age Treated With Oseltamivir; Test type: Superiority or Other; p = 0.008, Pairwise Wilcoxon
Statistical Analysis 3: Comparison: Children ≤5 Years of Age Treated With Oseltamivir vs Adults Treated With Oseltamivir; Test type: Superiority or Other; p < 0.0001, Pairwise Wilcoxon

14. Secondary Outcome: Time to Non-Detection of Viral RNA Among Participants With Influenza B Infections
Description: as for outcome 11
Time Frame: From Baseline (Day 1) to Day 10 (assessed on Days 1, 3, 6, 10)
Population: ALCIP Population. The "Number of Participants Analyzed" reflects the number of participants with influenza B infection who provided sufficient post-Baseline data.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Children ≤5 Years of Age Treated With Oseltamivir | Children 6 to 12 Years of Age Treated With Oseltamivir | Adults Treated With Oseltamivir
Number analyzed (Participants) | 130 | 199 | 207
days | 9.8 [8.1 to 10.1] | 10.0 [8.9 to 10.2] | 7.4 [6.9 to 7.9]
Statistical Analysis 1: Comparison: Children ≤5 Years of Age Treated With Oseltamivir vs Children 6 to 12 Years of Age Treated With Oseltamivir vs Adults Treated With Oseltamivir; Test type: Superiority or Other; p = 0.0002, Kruskal-Wallis
Statistical Analysis 2: Comparison: Children ≤5 Years of Age Treated With Oseltamivir vs Adults Treated With Oseltamivir; Test type: Superiority or Other; p = 0.008, Pairwise Wilcoxon
Statistical Analysis 3: Comparison: Children 6 to 12 Years of Age Treated With Oseltamivir vs Adults Treated With Oseltamivir; Test type: Superiority or Other; p < 0.0001, Pairwise Wilcoxon

15. Secondary Outcome: Viral Load Among Adults Treated With Oseltamivir
Description: Viral load was determined for those with detectable virus above the lower limit of quantification (LLQ) of 1.82 for influenza A viruses and 1.99 for influenza B viruses. The viral load from each sample was averaged among all participants and expressed in log10 of the number of viral particles per milliliter (log10 vp/mL).
Time Frame: Days 1, 3, 6, 10
Population: ALCIP Population. The "Number of Participants Analyzed" reflects the highest total number of participants who provided evaluable data for their viral RNA subtype at any visit. The number of participants who provided evaluable data for each viral RNA subtype at the specified visit (n) is shown in the table.
Measure: Mean (Standard Deviation); unit: log10 vp/mL
Arm/Group | Adults Treated With Oseltamivir
Number analyzed (Participants) | 959
log10 vp/mL
  Day 1, Total (n=959) | 5.8 (1.18)
  Day 1, H1N1 Seasonal (n=12) | 5.7 (1.22)
  Day 1, H3N2 (n=417) | 5.8 (1.23)
  Day 1, H1N1pdm09 (n=323) | 5.7 (1.15)
  Day 1, Influenza B (n=207) | 5.9 (1.09)
  Day 3, Total (n=781) | 4.2 (1.17)
  Day 3, H1N1 Seasonal (n=10) | 4.2 (1.34)
  Day 3, H3N2 (n=341) | 3.9 (1.15)
  Day 3, H1N1pdm09 (n=258) | 4.1 (1.07)
  Day 3, Influenza B (n=172) | 4.7 (1.19)
  Day 6, Total (n=317) | 3.3 (1.05)
  Day 6, H1N1 Seasonal (n=4) | 4.1 (0.48)
  Day 6, H3N2 (n=144) | 3.2 (1.06)
  Day 6, H1N1pdm09 (n=110) | 3.1 (0.93)
  Day 6, Influenza B (n=59) | 3.9 (1.04)
  Day 10, Total (n=88) | 3.0 (0.88)
  Day 10, H3N2 (n=44) | 2.9 (0.87)
  Day 10, H1N1pdm09 (n=33) | 2.8 (0.79)
  Day 10, Influenza B (n=11) | 3.7 (0.84)

16. Secondary Outcome: Viral Load Among Children Treated With Oseltamivir
Description: Viral load was determined for those with detectable virus above the LLQ of 1.82 for influenza A viruses and 1.99 for influenza B viruses. The viral load from each sample was averaged among all participants and expressed in log10 vp/mL.
Time Frame: Days 1, 3, 6, 10
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: log10 vp/mL
Arm/Group | Children Treated With Oseltamivir
Number analyzed (Participants) | 1283
log10 vp/mL
  Day 1, Total (n=1283) | 5.8 (1.15)
  Day 1, H3N2 (n=583) | 5.6 (1.22)
  Day 1, H1N1pdm09 (n=371) | 5.7 (1.13)
  Day 1, Influenza B (n=329) | 6.1 (0.98)
  Day 3, Total (n=1050) | 4.5 (1.25)
  Day 3, H3N2 (n=453) | 4.1 (1.16)
  Day 3, H1N1pdm09 (n=315) | 4.3 (1.12)
  Day 3, Influenza B (n=282) | 5.2 (1.19)
  Day 6, Total (n=628) | 3.8 (1.18)
  Day 6, H3N2 (n=271) | 3.6 (1.19)
  Day 6, H1N1pdm09 (n=181) | 3.7 (1.21)
  Day 6, Influenza B (n=176) | 4.1 (1.08)
  Day 10, Total (n=197) | 3.3 (0.99)
  Day 10, H3N2 (n=73) | 3.1 (1.01)
  Day 10, H1N1pdm09 (n=64) | 3.1 (0.84)
  Day 10, Influenza B (n=60) | 3.6 (1.04)

17. Secondary Outcome: Percentage of Participants With Symptom Resolution on Day 6 Comparing Resistant and Susceptible Viruses
Description: Pre-defined mutations in viral RNA were noted, the presence of which was defined as genotypic resistance. Phenotypic resistance was defined as 50% inhibitory concentration (IC50) more than 10-fold higher than the median value for all viruses of the same subtype. Treatment-emergent resistance was defined as the presence of genotypic or phenotypic resistance from a post-Baseline sample in the setting of a previously non-resistant Baseline sample. Susceptible viruses were those that did not exhibit treatment-emergent resistance. The percentage of participants with mild or absent symptoms on Day 6 was reported and stratified by resistant and susceptible viruses.
Time Frame: Day 6
Population: ALCIP Population. The "Number of Participants Analyzed" reflects the total number of participants with wild-type infection status at Baseline who provided evaluable data at the Day 6 visit. The number of participants who provided evaluable data for each resistance status at the Day 6 visit (n) is shown in the table.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Treated With Oseltamivir
Number analyzed (Participants) | 1730
percentage of participants
  Total (n=1730) | 61.2
  Resistant (n=59) | 55.9
  Susceptible (n=1671) | 61.4
Statistical Analysis 1: Comparison: Participants Treated With Oseltamivir; Resistant versus Susceptible; Test type: Superiority or Other; p = 0.4464, Cochran-Mantel-Haenszel

18. Secondary Outcome: Percentage of Participants by Day of Viral RNA First Not Detected Comparing Resistant and Susceptible Viruses
Description: Pre-defined mutations in viral RNA were noted, the presence of which was defined as genotypic resistance. Phenotypic resistance was defined as IC50 more than 10-fold higher than the median value for all viruses of the same subtype. Treatment-emergent resistance was defined as the presence of genotypic or phenotypic resistance from a post-Baseline sample in the setting of a previously non-resistant Baseline sample. Susceptible viruses were those that did not exhibit treatment-emergent resistance. The percentage of participants by earliest post-Baseline test day on which viral RNA was not detected was reported and stratified by resistant and susceptible viruses.
Time Frame: Days 3, 6, 10
Population: ALCIP Population. The "Number of Participants Analyzed" reflects the total number of participants with wild-type infection status at Baseline who provided evaluable data at the specified visit. The number of participants who provided evaluable data for each resistance status at the specified visit (n) is shown in the table.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Treated With Oseltamivir
Number analyzed (Participants) | 1682
percentage of participants
  Day 3, Total (n=1682) | 15.3
  Day 3, Resistant (n=59) | 0
  Day 3, Susceptible (n=1623) | 15.8
  Day 6, Total (n=1682) | 40.5
  Day 6, Resistant (n=59) | 10.2
  Day 6, Susceptible (n=1623) | 41.7
  Day 10, Total (n=1682) | 30.4
  Day 10, Resistant (n=59) | 59.3
  Day 10, Susceptible (n=1623) | 29.4
Statistical Analysis 1: Comparison: Participants Treated With Oseltamivir; Resistant versus Susceptible; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel

19. Secondary Outcome: Percentage of Participants With Resistant Versus Susceptible Viruses by Baseline Viral Load
Description: Pre-defined mutations in viral RNA were noted, the presence of which was defined as genotypic resistance. Phenotypic resistance was defined as IC50 more than 10-fold higher than the median value for all viruses of the same subtype. Treatment-emergent resistance was defined as the presence of genotypic or phenotypic resistance from a post-Baseline sample in the setting of a previously non-resistant Baseline sample. Susceptible viruses were those that did not exhibit treatment-emergent resistance. The mean viral load from each sample was expressed in log10 vp/mL and stratified by resistant and susceptible viruses.
Time Frame: Baseline (Day 1)
Population: ALCIP Population. The "Number of Participants Analyzed" reflects the total number of participants with wild-type infection status at Baseline who provided evaluable data. The number of participants who provided evaluable data for each resistance status at Baseline (n) is shown in the table.
Measure: Number; unit: percentage of participants
Arm/Group | Participants Treated With Oseltamivir
Number analyzed (Participants) | 1802
percentage of participants
  Total, Resistant (n=1802) | 3.2
  Total, Susceptible (n=1802) | 96.8
  Viral Load <4.95, Resistant (n=452) | 2.0
  Viral Load <4.95, Susceptible (n=452) | 98.0
  Viral Load 4.95 to 5.89, Resistant (n=450) | 3.8
  Viral Load 4.95 to 5.89, Susceptible (n=450) | 96.2
  Viral Load 5.89 to 6.61, Resistant (n=457) | 3.1
  Viral Load 5.89 to 6.61, Susceptible (n=457) | 96.9
  Viral Load >6.61, Resistant (n=443) | 3.8
  Viral Load >6.61, Susceptible (n=443) | 96.2
Statistical Analysis 1: Comparison: Participants Treated With Oseltamivir; Resistant versus Susceptible; Test type: Superiority or Other; p = 0.2499, Cochran-Mantel-Haenszel

20. Secondary Outcome: Total Daily Symptom Score According to Global Assessment by the Investigator Among Adults Treated With Oseltamivir
Description: Symptoms were assessed on Days 1, 6, and 10. The Investigator rated seven symptoms of fever, sore throat, nasal congestion, cough, aches/pains, headache, and fatigue on a scale of 0 (absent/no problem) to 3 (severe/major problem). The global score was calculated as a sum of all individual symptom scores. Global scores may range from 0 to 21, with higher scores indicating worse or more pronounced symptoms.
Time Frame: Days 1, 6, 10
Population: ALCIP Population. The "Number of Participants Analyzed" reflects the total number of participants who provided evaluable data for their viral RNA subtype at the specified visit. The number of participants who provided evaluable data for each viral RNA subtype at the specified visit (n) is shown in the table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adults Treated With Oseltamivir
Number analyzed (Participants) | 961
units on a scale
  Day 1, Total (n=960) | 12.3 (5.03)
  Day 1, H1N1 Seasonal (n=12) | 11.4 (6.02)
  Day 1, H3N2 (n=419) | 11.2 (5.41)
  Day 1, H1N1pdm09 (n=323) | 13.2 (4.28)
  Day 1, Influenza B (n=206) | 13.4 (4.76)
  Day 6, Total (n=890) | 3.7 (3.27)
  Day 6, H1N1 Seasonal (n=9) | 2.8 (2.91)
  Day 6, H3N2 (n=383) | 3.4 (3.03)
  Day 6, H1N1pdm09 (n=307) | 3.8 (3.28)
  Day 6, Influenza B (n=191) | 4.1 (3.66)
  Day 10, Total (n=827) | 2.0 (2.51)
  Day 10, H3N2 (n=357) | 2.1 (2.6)
  Day 10, H1N1pdm09 (n=281) | 1.9 (2.36)
  Day 10, Influenza B (n=189) | 2.1 (2.57)

21. Secondary Outcome: Total Daily Symptom Score According to Global Assessment by the Investigator Among Children Treated With Oseltamivir
Description: Symptoms were assessed on Days 1, 6, and 10. The Investigator rated seven symptoms of fever, sore throat, nasal congestion, cough, aches/pains, headache, and energy/tiredness on a scale of 0 (absent/no problem) to 3 (severe/major problem). The global score was calculated as a sum of all individual symptom scores. Global scores may range from 0 to 21, with higher scores indicating worse or more pronounced symptoms.
Time Frame: Days 1, 6, 10
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Children Treated With Oseltamivir
Number analyzed (Participants) | 1283
units on a scale
  Day 1, Total (n=1283) | 12.4 (3.92)
  Day 1, H3N2 (n=583) | 12.3 (3.77)
  Day 1, H1N1pdm09 (n=371) | 11.9 (4.02)
  Day 1, Influenza B (n=329) | 13.0 (3.98)
  Day 6, Total (n=1252) | 3.3 (2.83)
  Day 6, H3N2 (n=567) | 3.2 (2.57)
  Day 6, H1N1pdm09 (n=364) | 3.2 (2.60)
  Day 6, Influenza B (n=321) | 3.5 (3.44)
  Day 10, Total (n=1228) | 1.3 (1.59)
  Day 10, H3N2 (n=562) | 1.3 (1.59)
  Day 10, H1N1pdm09 (n=350) | 1.4 (1.54)
  Day 10, Influenza B (n=316) | 1.3 (1.63)

22. Secondary Outcome: Body Temperature Among Adults Treated With Oseltamivir
Description: Body temperature was measured by the Investigator using an oral or tympanic thermometer at Baseline and Day 10. Body temperature at each visit was averaged among all participants and expressed in degrees Celsius.
Time Frame: Days 1, 10
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Adults Treated With Oseltamivir
Number analyzed (Participants) | 960
degrees Celsius
  Day 1, Total (n=960) | 38.0 (0.91)
  Day 1, H1N1 Seasonal (n=12) | 37.8 (1.10)
  Day 1, H3N2 (n=418) | 37.8 (0.89)
  Day 1, H1N1pdm09 (n=323) | 38.2 (0.88)
  Day 1, Influenza B (n=207) | 38.0 (0.90)
  Day 10, Total (n=827) | 36.6 (0.40)
  Day 10, H3N2 (n=356) | 36.6 (0.40)
  Day 10, H1N1pdm09 (n=282) | 36.6 (0.38)
  Day 10, Influenza B (n=189) | 36.6 (0.41)

23. Secondary Outcome: Change From Baseline in Body Temperature Among Adults Treated With Oseltamivir
Description: Body temperature was measured by the Investigator using an oral or tympanic thermometer at Baseline and Day 10. The change in body temperature between visits was averaged among all participants and expressed in degrees Celsius.
Time Frame: Baseline (Day 1) to Day 10
Population: ALCIP Population. The "Number of Participants Analyzed" reflects the total number of participants who provided evaluable data for their viral RNA subtype at Baseline and Day 10. The number of participants who provided evaluable data for each viral RNA subtype at Baseline and Day 10 (n) is shown in the table.
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Adults Treated With Oseltamivir
Number analyzed (Participants) | 826
degrees Celsius
  Total (n=826) | -1.4 (0.96)
  H3N2 (n=355) | -1.2 (0.94)
  H1N1pdm09 (n=282) | -1.7 (0.93)
  Influenza B (n=189) | -1.4 (0.95)

24. Secondary Outcome: Body Temperature Among Children Treated With Oseltamivir
Description: as for outcome 22
Time Frame: Days 1, 10
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Children Treated With Oseltamivir
Number analyzed (Participants) | 1282
degrees Celsius
  Day 1, Total (n=1282) | 38.3 (0.93)
  Day 1, H3N2 (n=583) | 38.3 (0.98)
  Day 1, H1N1pdm09 (n=370) | 38.3 (0.91)
  Day 1, Influenza B (n=329) | 38.2 (0.87)
  Day 10, Total (n=1223) | 36.7 (0.38)
  Day 10, H3N2 (n=560) | 36.6 (0.37)
  Day 10, H1N1pdm09 (n=346) | 36.7 (0.40)
  Day 10, Influenza B (n=317) | 36.6 (0.38)

25. Secondary Outcome: Change From Baseline in Body Temperature Among Children Treated With Oseltamivir
Description: as for outcome 23
Time Frame: Baseline (Day 1) to Day 10
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Children Treated With Oseltamivir
Number analyzed (Participants) | 1222
degrees Celsius
  Total (n=1222) | -1.6 (0.98)
  H3N2 (n=560) | -1.6 (1.02)
  H1N1pdm09 (n=345) | -1.5 (0.97)
  Influenza B (n=317) | -1.6 (0.91)

ADVERSE EVENTS:
Time Frame: From Baseline (Day 1) to Day 10; assessed on Days 1, 3, 6, 10
Description: AEHP Population.
Groups:
- Participants Not Treated With Oseltamivir: Otherwise healthy/non-immunocompromised adults and children with a positive diagnostic test of influenza and/or displaying symptoms suggestive of influenza-like illness were enrolled during Years 1 to 7 of the overall study. Participants not receiving oseltamivir, including no treatment or other antiviral treatment, were followed for up to 10 days after informed consent for virological surveillance and assessment of clinical outcomes.
Arm/Group | Participants Treated With Oseltamivir | Participants Not Treated With Oseltamivir
Serious Adverse Events (participants affected / at risk) | 24/2578 | 11/1975
Other Adverse Events (participants affected / at risk) | 0/2578 | 0/1975
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants Treated With Oseltamivir (N=2578) | Participants Not Treated With Oseltamivir (N=1975)
Pneumonia (Infections and infestations) | 5 | 1
Bronchitis (Infections and infestations) | 0 | 2
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Scarlet fever (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1

LIMITATIONS AND CAVEATS:
This was a non-randomized, observational study and many comparisons were not powered to detect a true statistically significant difference between groups. Inferential analyses should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.